CLINICAL TRIAL: NCT03626051
Title: Effects of Rigid Ankle Tape and Fibular Tape on Functional Performance in Participants With Functional Ankle Instability
Brief Title: Ankle Taping and Functional Ankle Instability
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: National Yang Ming Chiao Tung University (Other)
Responsible Party: Principal Investigator, Yea-Ru Yang, Professor, National Yang Ming Chiao Tung University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: YM106003F
Record Dates: First submitted 2017-04-06; First posted 2018-08-10 (Actual); Last update posted 2018-08-10 (Actual); Status verified 2018-08

CONDITIONS: Ankle Sprains
Keywords: ankle taping
MeSH Terms: conditions — Ankle Injuries

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- rigid tape group (Active Comparator)
  Interventions: Device: Rigid tape
- fibular tape group (Experimental)
  Interventions: Device: Fibular tape

INTERVENTIONS:
Device: Rigid tape — This taping method used an anchor, two stirrups, three figure-six's (two preventing inversion and one preventing eversion), heel lock and a lock off. Adhesive rigid strapping tape (Leuko Sports Tape, Beiersdorf Australia Ltd, North Ryde) of 3.8 cm thickness was used for all participants
  Arms: rigid tape group
Device: Fibular tape — This taping method used a rigid strapping tape to reinforce a posterior-superior mobilisation of the distal fibula. Tension was applied on the tape in a posterior and superior direction. Adhesive rigid strapping tape (Leuko Sports Tape, Beiersdorf Australia Ltd, North Ryde) of 3.8 cm thickness was used for all participants
  Arms: fibular tape group

SUMMARY:
Background and purpose:

Ankle inversion sprains are the commonest injuries of the lower extremities. Taping is routinely used after ankle sprain to support the joint and prevent reinjury. The effect of taping on functional performance in participants after ankle sprain has received little attention and generally with inconsistent findings. Besides, the perception of confidence and reassurance that may come with the ankle being taped might lead to the improvement of functional mobility performance. Therefore, the purpose of this study is to investigate the effects of rigid ankle tape and fibular tape on functional performance, self-efficacy and perceived stability, confidence and reassurance during functional tasks in participants with functional ankle instability.

Methods:

This study is a randomized controlled trial. Forty subjects with functional ankle instability will be recruited and randomly assigned into the rigid tape group and the fibular tape group. Participants will perform functional mobility tests with and without the ankle taped. The functional tests are: figure-8 hopping test, lateral hopping test, star excursion balance test (SEBT), single-leg stance and stair decent test. Secondary outcome measures were self-efficacy and perception measure.

Statistics:

Two-way analysis of variance with repeated measures was used to determine the effects of intervention on each dependent variable. Model effects were group, time (pre, post), and their interaction. Post hoc pairwise comparisons between pre and post in each group, and independent t test between groups, were used to document the difference. The statistical significance was set at p less than 0.05.

ELIGIBILITY:
Inclusion Criteria:

1. participants had to have sustained at least two ankle sprain from a sudden inversion trauma, at least one month prior, which resulted in pain and swelling over the lateral ligament and limping, and have at least moderate functional ankle instability
2. a score of <27 on the Cumberland Ankle Instability Tool (CAIT)
3. anterior drawer test: negative
4. talar tilt test: negative

Exclusion Criteria:

1. if they had sprained their ankle within two weeks of testing
2. had a neurological or vestibular disorder or were unable to understand the nature of the protocol and test instructions.
3. have received intervention for ankle instability
4. PI's research assistant -

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2017-04-06 (Actual); Primary Completion 2017-05-29 (Actual); Study Completion 2017-06-27 (Actual)

PRIMARY OUTCOMES:
Figure-8 hopping test | Change from baseline at one hour
  This test consists of hopping twice around a 5 m course on the test foot in a figure-8, as quickly as possible. The time taken for the participant to complete two circuits of the figure-8 was measured using a stopwatch, and the average of the two best times out of three attempts was recorded.
Lateral hopping test | Change from baseline at one hour
  participants were instructed to hop laterally 30 cm and back for a total of 10 repetitions. The total time was recorded with a handheld stopwatch to the nearest 0.01 second.
Star excursion balance test | Change from baseline at one hour
  This test examined the ability to balance on the affected leg while reaching in various directions with the other foot. Participants stood on the test foot at the central point, and using the other foot reached as far as possible in each of three of the 8 directions of the star excursion balance test (anterior, posterior and postero-medial, relative to the test foot). Only three directions were used due to redundancy among the eight directions. Participants made three attempts in each test direction with the average of the best two attempts for each direction recorded in centimetre
Single-leg stance test | Change from baseline at one hour
  Participants were instructed to balance on one leg for 30 s with their eyes closed, arms at their side, and the other foot touching the medial side of the supporting calf. If they lost their balance, participants were instructed to keep their eyes closed and attempt to re-establish their balance. The number of foot movements made by the stance foot during the 30 s was counted. A foot movement was counted if any of the following occurred: loss of contact with the ground by any part of the foot; a change in foot direction; or each instance when the contralateral foot touched the ground. The lowest total number of foot movements from three attempts was recorded.
Stair decent test | Change from baseline at one hour
  Participants were instructed to run down a flight of 11 stairs as quickly as possible, ensuring that they made contact with every step with one foot, and without using the handrail.The time taken from the first step to touchdown by both feet at the bottom of the flight of stairs was measured. The two best times out of three attempts was averaged.

SECONDARY OUTCOMES:
Self-efficacy questionnaire | Change from baseline at one hour
  The self-efficacy questionnaire was modified from the pain self-efficacy questionnaire, to compare participants' self-reported confidence in performing a range of functionally challenging tasks. The questionnaire consisted of 17 items related to tasks of increasing difficulty. Participants rated their level of confidence in their ability to perform each activity.
Self-perception measure | Change from baseline at one hour
  Three perception measures were recorded at the completion of each functional test to determine whether there was a difference in participants' perceptions between the tape and no tape conditions. Participants recorded their perception of ankle stability, confidence and reassurance. Stability was defined as "how stable your ankle felt during the test", confidence as "how positive you felt during the test", and reassurance as "how safe you felt during the test".

CONTACTS AND LOCATIONS:
Locations (1):
- National Yang-Ming University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Result] Handoll HH, Rowe BH, Quinn KM, de Bie R. Interventions for preventing ankle ligament injuries. Cochrane Database Syst Rev. 2001;(3):CD000018. doi: 10.1002/14651858.CD000018. PMID 11686947
- [Result] Cordova ML, Ingersoll CD, LeBlanc MJ. Influence of ankle support on joint range of motion before and after exercise: a meta-analysis. J Orthop Sports Phys Ther. 2000 Apr;30(4):170-7; discussion 178-82. doi: 10.2519/jospt.2000.30.4.170. PMID 10778794
- [Result] Abian-Vicen J, Alegre LM, Fernandez-Rodriguez JM, Aguado X. Prophylactic ankle taping: elastic versus inelastic taping. Foot Ankle Int. 2009 Mar;30(3):218-25. doi: 10.3113/FAI.2009.0218. PMID 19321098
- [Result] Broglio SP, Monk A, Sopiarz K, Cooper ER. The influence of ankle support on postural control. J Sci Med Sport. 2009 May;12(3):388-92. doi: 10.1016/j.jsams.2007.12.010. Epub 2008 Jun 11. PMID 18550434
- [Result] Meana M, Alegre LM, Elvira JL, Aguado X. Kinematics of ankle taping after a training session. Int J Sports Med. 2008 Jan;29(1):70-6. doi: 10.1055/s-2007-965126. Epub 2007 Jul 5. PMID 17614032
- [Result] MacKean LC, Bell G, Burnham RS. Prophylactic ankle bracing vs. taping: effects on functional performance in female basketball players. J Orthop Sports Phys Ther. 1995 Aug;22(2):77-81. doi: 10.2519/jospt.1995.22.2.77. PMID 7581435
- [Result] Verbrugge JD. The effects of semirigid Air-Stirrup bracing vs. adhesive ankle taping on motor performance. J Orthop Sports Phys Ther. 1996 May;23(5):320-5. doi: 10.2519/jospt.1996.23.5.320. PMID 8728530
- [Result] Burks RT, Bean BG, Marcus R, Barker HB. Analysis of athletic performance with prophylactic ankle devices. Am J Sports Med. 1991 Mar-Apr;19(2):104-6. doi: 10.1177/036354659101900202. PMID 2039059
- [Result] Jerosch J, Thorwesten L, Frebel T, Linnenbecker S. Influence of external stabilizing devices of the ankle on sport-specific capabilities. Knee Surg Sports Traumatol Arthrosc. 1997;5(1):50-7. doi: 10.1007/s001670050025. PMID 9127855
- [Result] Paris DL. The Effects of the Swede-O, New Cross, and McDavid Ankle Braces and Adhesive Ankle Taping on Speed, Balance, Agility, and Vertical Jump. J Athl Train. 1992;27(3):253-6. PMID 16558170
- [Result] Sawkins K, Refshauge K, Kilbreath S, Raymond J. The placebo effect of ankle taping in ankle instability. Med Sci Sports Exerc. 2007 May;39(5):781-7. doi: 10.1249/MSS.0b013e3180337371. PMID 17468574
- [Result] Moiler K, Hall T, Robinson K. The role of fibular tape in the prevention of ankle injury in basketball: A pilot study. J Orthop Sports Phys Ther. 2006 Sep;36(9):661-8. doi: 10.2519/jospt.2006.2259. PMID 17017271
- [Result] Gutierrez GM, Kaminski TW, Douex AT. Neuromuscular control and ankle instability. PM R. 2009 Apr;1(4):359-65. doi: 10.1016/j.pmrj.2009.01.013. PMID 19627919
- [Result] Hubbard TJ. Ligament laxity following inversion injury with and without chronic ankle instability. Foot Ankle Int. 2008 Mar;29(3):305-11. doi: 10.3113/FAI.2008.0305. PMID 18348827
- [Result] Hoch MC, Staton GS, Medina McKeon JM, Mattacola CG, McKeon PO. Dorsiflexion and dynamic postural control deficits are present in those with chronic ankle instability. J Sci Med Sport. 2012 Nov;15(6):574-9. doi: 10.1016/j.jsams.2012.02.009. Epub 2012 May 8. PMID 22575498
- [Result] Denegar CR, Hertel J, Fonseca J. The effect of lateral ankle sprain on dorsiflexion range of motion, posterior talar glide, and joint laxity. J Orthop Sports Phys Ther. 2002 Apr;32(4):166-73. doi: 10.2519/jospt.2002.32.4.166. PMID 11949665
- [Result] Whitman JM, Cleland JA, Mintken PE, Keirns M, Bieniek ML, Albin SR, Magel J, McPoil TG. Predicting short-term response to thrust and nonthrust manipulation and exercise in patients post inversion ankle sprain. J Orthop Sports Phys Ther. 2009 Mar;39(3):188-200. doi: 10.2519/jospt.2009.2940. PMID 19252260
- [Result] Wikstrom EA, Hubbard TJ. Talar positional fault in persons with chronic ankle instability. Arch Phys Med Rehabil. 2010 Aug;91(8):1267-71. doi: 10.1016/j.apmr.2010.04.022. PMID 20684909
- [Result] Hopkins JT, Brown TN, Christensen L, Palmieri-Smith RM. Deficits in peroneal latency and electromechanical delay in patients with functional ankle instability. J Orthop Res. 2009 Dec;27(12):1541-6. doi: 10.1002/jor.20934. PMID 19569189
- [Result] Munn J, Sullivan SJ, Schneiders AG. Evidence of sensorimotor deficits in functional ankle instability: a systematic review with meta-analysis. J Sci Med Sport. 2010 Jan;13(1):2-12. doi: 10.1016/j.jsams.2009.03.004. Epub 2009 May 12. PMID 19442581
- [Result] Van Deun S, Staes FF, Stappaerts KH, Janssens L, Levin O, Peers KK. Relationship of chronic ankle instability to muscle activation patterns during the transition from double-leg to single-leg stance. Am J Sports Med. 2007 Feb;35(2):274-81. doi: 10.1177/0363546506294470. Epub 2006 Dec 27. PMID 17192320
- [Result] Mitchell A, Dyson R, Hale T, Abraham C. Biomechanics of ankle instability. Part 1: Reaction time to simulated ankle sprain. Med Sci Sports Exerc. 2008 Aug;40(8):1515-21. doi: 10.1249/mss.0b013e31817356b6. PMID 18705024
- [Result] Mitchell A, Dyson R, Hale T, Abraham C. Biomechanics of ankle instability. Part 2: Postural sway-reaction time relationship. Med Sci Sports Exerc. 2008 Aug;40(8):1522-8. doi: 10.1249/MSS.0b013e31817356d6. PMID 18614937
- [Result] Bicici S, Karatas N, Baltaci G. Effect of athletic taping and kinesiotaping(R) on measurements of functional performance in basketball players with chronic inversion ankle sprains. Int J Sports Phys Ther. 2012 Apr;7(2):154-66. PMID 22530190
- [Result] Delahunt E, McGrath A, Doran N, Coughlan GF. Effect of taping on actual and perceived dynamic postural stability in persons with chronic ankle instability. Arch Phys Med Rehabil. 2010 Sep;91(9):1383-9. doi: 10.1016/j.apmr.2010.06.023. PMID 20801256
- [Result] Halim-Kertanegara S, Raymond J, Hiller CE, Kilbreath SL, Refshauge KM. The effect of ankle taping on functional performance in participants with functional ankle instability. Phys Ther Sport. 2017 Jan;23:162-167. doi: 10.1016/j.ptsp.2016.03.005. Epub 2016 Apr 18. PMID 27262625
- [Result] Hiller CE, Refshauge KM, Bundy AC, Herbert RD, Kilbreath SL. The Cumberland ankle instability tool: a report of validity and reliability testing. Arch Phys Med Rehabil. 2006 Sep;87(9):1235-41. doi: 10.1016/j.apmr.2006.05.022. PMID 16935061
- [Result] Docherty CL, Arnold BL, Gansneder BM, Hurwitz S, Gieck J. Functional-Performance Deficits in Volunteers With Functional Ankle Instability. J Athl Train. 2005 Mar;40(1):30-34. PMID 15902321
- [Result] Munro AG, Herrington LC. Between-session reliability of the star excursion balance test. Phys Ther Sport. 2010 Nov;11(4):128-32. doi: 10.1016/j.ptsp.2010.07.002. Epub 2010 Aug 17. PMID 21055706
- [Result] Olmsted LC, Carcia CR, Hertel J, Shultz SJ. Efficacy of the Star Excursion Balance Tests in Detecting Reach Deficits in Subjects With Chronic Ankle Instability. J Athl Train. 2002 Dec;37(4):501-506. PMID 12937574
- [Result] Hiller CE, Refshauge KM, Herbert RD, Kilbreath SL. Balance and recovery from a perturbation are impaired in people with functional ankle instability. Clin J Sport Med. 2007 Jul;17(4):269-75. doi: 10.1097/JSM.0b013e3180f60b12. PMID 17620780
- [Result] Hiller CE, Refshauge KM, Herbert RD, Kilbreath SL. Intrinsic predictors of lateral ankle sprain in adolescent dancers: a prospective cohort study. Clin J Sport Med. 2008 Jan;18(1):44-8. doi: 10.1097/JSM.0b013e31815f2b35. PMID 18185038